CLINICAL TRIAL: NCT02548117
Title: H-36371: Finasteride as a Method of Managing Testosterone-Induced Erythrocytosis
Brief Title: H-36731: Finasteride in Management of Elevated Red Blood Cells
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding was not available.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Larry I. Lipshultz, Professor of Urology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-15-40-10
Record Dates: First submitted 2015-09-02; First posted 2015-09-14 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: ERYTHROCYTOSIS
Keywords: Testosterone therapy; erythrocytosis; finasteride
MeSH Terms: conditions — Polycythemia | interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride (Active Comparator): ARM 1 subjects will receive finasteride 5 mg orally daily.
  Interventions: Drug: Finasteride
- No Treatment (No Intervention): The ARM 2 (control group) will not receive any study treatment.

INTERVENTIONS:
Drug: Finasteride — Subjects will take 5 mg finasteride orally every day for about 2 years.
  Other Names: Proscar
  Arms: Finasteride

SUMMARY:
Hypogonadism (low testosterone) is becoming an increasingly recognized problem that affects numerous men in the United States. Symptoms may be always feeling tired, lower sex drive, and loss of muscle mass. Treatment typically involves testosterone in either injections or a topical gel form.

However, administration of testosterone is not without side effects of its own. Testosterone supplementation therapy is known to cause a variety of side effects including high blood pressure and high lipids (fats) and an increased proportion of red blood cells. Side effects of increased red blood cells can include an increased risk of developing a blood clot.

The increase in the red blood cells is related to dihydrotestosterone (DHT - a male sex hormone) activity. It is normal for the testosterone to become DHT. DHT has various effects on the body including growth of the prostate gland, baldness, and others and DHT levels have been linked to elevated red blood cell counts in men on testosterone.

Finasteride is an FDA approved medication used in the treatment of benign prostatic hypertrophy (BPH) in men with enlarged prostate to improve symptoms and to reduce the risk of the need for surgery. Finasteride may prevent elevations in or reduce elevated red blood cell levels in men on testosterone.

DETAILED DESCRIPTION:
Hypogonadism is becoming an increasingly recognized clinical syndrome affecting millions of men in the United States and globally, and is characterized by symptoms including chronic fatigue, decreased libido and muscle mass, and low serum testosterone level. Treatment of hypogonadism in men typically involves treatment with exogenous testosterone.

However, exogenous testosterone therapy is not without risks, and can cause numerous side effects including high blood pressure, hyperlipidemia, and erythrocytosis, or elevated hematocrit. Adverse effects of erythrocytosis can include an increased risk of developing thromboembolism, and treatment of erythrocytosis involves therapeutic phlebotomy and testosterone dose adjustment, which can decrease the symptomatic benefits of testosterone therapy.

Aghazadeh et al.found that erythrocytosis occurring during testosterone therapy may be related to dihydrotestosterone (DHT) levels. As part of normal physiology, testosterone is converted to DHT via 5-alpha reductase (5AR). DHT is associated with various effects on the body, including stimulation of prostate growth, male pattern baldness, and others. Currently, finasteride, a 5-alpha reductase inhibitor (5ARI), is available as an FDA-approved drug used to treat DHT-related prostate growth and to prevent DHT-related baldness.

Given the positive association between DHT and the increased hematocrit seen in men being treated for hypogonadism with exogenous testosterone, finasteride's effects in preventing the synthesis of DHT may improve or even prevent erythrocytosis in men on testosterone.

The study will be a prospective randomized controlled trial of patients on injectable testosterone therapy. Subjects will be evenly distributed between the control and treatment groups. The treatment groups will receive finasteride and the control groups will not. All subjects will then be followed with blood tests to determine if there are any changes in their hematocrit, testosterone, DHT, and other blood test values.

An interim data analysis will be performed after approximately 150 men (75 treatment and 75 control) are accrued into the study and followed for at least 1 year. Rates of hematocrit elevation and erythrocytosis will be evaluated in finasteride treated and untreated men to determine whether finasteride is having an impact on erythrocytosis rates and whether any unanticipated adverse effects are occurring. Secondary outcomes, including effects on erythropoietin and hepcidin levels, will also be evaluated. Study accrual will continue if there is evidence that finasteride may decrease the incidence of erythrocytosis. The study will be stopped if unacceptable adverse events are identified or if there is no evidence suggesting that finasteride mitigates the risk of erythrocytosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 years of age or older
* Currently is being treated for hypogonadism with testosterone therapy using injectable testosterone.
* Must not have erythrocytosis (defined as a hematocrit of 52% or higher) attributable to other medication or medical condition
* Agree not to initiate any other treatment for erectile dysfunction (ED), including herbal and over- the-counter (OTC) medications, for the duration of the study.
* Must not already be taking finasteride or other 5-alpha reductase inhibitor

Exclusion Criteria:

* Men not currently using testosterone supplementation therapy or men on non-injectable testosterone therapy
* Prior history of anabolic steroid use, but have not used for at least 6 months
* Prior history of testosterone use, but have not used for at least 6 months
* Men who are already taking finasteride
* Untreated or inadequately treated hypothyroidism
* Significant history of allergy and/or sensitivity to the drug products or excipients, including sensitivity to testosterone and/or finasteride
* Current use of any medications, herbal, and/or nutritional supplements that can interfere with testosterone level
* Currently receiving treatment with cancer chemotherapy or anti-androgens
* Any contraindication to testosterone therapy or finasteride
* History of luteinizing hormone-releasing hormone antagonist or agonist treatment
* History of clomiphene treatment in 6 months prior to Visit 1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of serum hemoglobin parameters as a function of serum DHT levels | Approximately 2 years
  Comparison between the two ARMS will be done to determine if administration of finasteride may prevent elevations in or reduce levels of hemoglobin/hematocrit.
Evaluation of serum hematocrit parameters as a function of serum DHT levels | Approximately 2 years
  Comparison between the two ARMS will be done to determine if administration of finasteride may prevent elevations in or reduce levels of hemoglobin/hematocrit.
Evaluation of serum hormone parameters as a function of serum DHT levels | Approximately 2 years
  Comparison between the two ARMS will be done to determine if administration of finasteride may prevent elevations in or reduce levels of hemoglobin/hematocrit.

CONTACTS AND LOCATIONS:
Overall Officials: Larry I. Lipshultz, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States